CLINICAL TRIAL: NCT06536491
Title: A Randomized, Controlled, Subject- and Evaluator-Masked, Phase 2 Clinical Trial Comparing EC-104 Intravitreal Implant to Ozurdex® for the Treatment of Diabetic Macular Edema (BETTIS-1)
Brief Title: EC-104 Intravitreal Implant for the Treatment of Diabetic Macular Edema
Acronym: BETTIS-1
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Eclipse Life Sciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EC104-CS-201
Record Dates: First submitted 2024-07-31; First posted 2024-08-05 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Diabetic Macular Edema
MeSH Terms: interventions — Dexamethasone

STUDY DESIGN:
Intervention Model Description: Computer generated equal randomization
Who Masked: Participant, Outcomes Assessor
Masking Description: Evaluators of efficacy study assessments will be masked. The injecting physician and the injection technician or clinical assistant preparing the IP for administration will be unmasked to the identity of the specific investigational product (IP)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- EC-104 high dose (Experimental): Intravitreal implant of fluocinolone acetonide
  Interventions: Drug: EC-104 high dose
- EC-104 low dose (Experimental): Intravitreal implant of fluocinolone acetonide
  Interventions: Drug: EC-104 low dose
- Dexamethasone intravitreal implant (Active Comparator): Marketed product
  Interventions: Drug: Dexamethasone intravitreal implant

INTERVENTIONS:
Drug: EC-104 high dose — Intravitreal injection
  Arms: EC-104 high dose
Drug: EC-104 low dose — Intravitreal injection
  Arms: EC-104 low dose
Drug: Dexamethasone intravitreal implant — Marketed product intravitreal injection
  Arms: Dexamethasone intravitreal implant

SUMMARY:
This is a prospective, randomized, subject- and evaluator-masked, Phase 2, multicenter study comparing the safety and efficacy of EC-104-6M high-dose (fluocinolone acetonide [FA] 0.14 mg) implant and EC-104-4M low-dose (FA 0.092 mg) implant to Ozurdex® (dexamethasone intravitreal (IVT) implant, 0.7 mg) in subjects with diabetic retinopathy (DR) and center-involving diabetic macular edema (DME), with prior suboptimal clinical response to IVT anti-VEGF therapy who have been previously treated with locally administered corticosteroids without a clinically significant rise in intraocular pressure (IOP).

DETAILED DESCRIPTION:
Approximately 75 subjects who meet entry criteria will be randomized 1:1:1 to EC-104-6M high-dose (FA 0.14 mg) implant or EC-104-4M low-dose (FA 0.092 mg) implant or Ozurdex® (dexamethasone IVT implant 0.7 mg), with the goal of achieving approximately 20 subjects per group with a positive therapeutic response in their study eyes, who are evaluable in the primary endpoint analysis to assess efficacy. Subjects with a positive therapeutic response at Week 4 will be included in the primary and secondary endpoint analyses to assess efficacy for "Time to recurrent disease." Subjects who do not achieve a positive therapeutic response will be classified as suboptimal responders. While suboptimal responders will not be included in the primary and the secondary endpoint analyses to assess efficacy for "Time to recurrent disease," they will remain in the study and will be followed prospectively, with inclusion in the remaining endpoints to assess efficacy and all safety endpoint analyses

ELIGIBILITY:
Inclusion Criteria:

1. Males or females who are at least 18 years of age at the time of informed consent
2. Willing and able to provide signed informed consent (participant or legally authorized representative) prior to any study-related procedures and to comply with all study visits and cooperate with all examinations
3. Diagnosis of diabetes mellitus (Type 1 or Type 2), with history of diabetic macular edema (DME) < = years duration prior to Screening Visit 1
4. Currently monitored hemoglobin A1c values ≤ 10.0 while under the care of a qualified medical provider for diabetes mellitus management, unless provider allows value variance

   Inclusion criteria for the study eye (all of the below criteria must be met in the same eye):
5. Early Treatment Diabetic Retinopathy Study BCVA score ≤ 70 letters (Snellen equivalent 20/40 or worse) and ≥ 20 letters (Snellen equivalent 20/400) in at least 1 eye

Exclusion Criteria:

1. Previous or current diagnosis of any form of glaucoma (defined as cup-to-disc ratio > 0.7) or ocular hypertension (documented intraocular pressure (IOP) > 21 mm Hg without glaucomatous disc damage) requiring medical or surgical intervention
2. History of steroid-induced IOP elevation > 25 mm Hg
3. Presence of active proliferative diabetic retinopathy, defined as active neovascularization of disc (NVD), neovascularization elsewhere (NVE), neovascularization of iris (NVI), neovascularization of angle (NVA), or vitreous hemorrhage in the setting of active NVD or NVE

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-08-19 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Ocular and Systemic Safety | Through Week 24
  Incidence of Adverse events

SECONDARY OUTCOMES:
Diabetic macular edema recurrence | Through Week 24
  Time (days) to recurrence

CONTACTS AND LOCATIONS:
Locations (1):
- Retina Associates of Florida, LLC, Tampa, Florida, United States

IPD SHARING:
Plan to Share IPD: No